CLINICAL TRIAL: NCT06064149
Title: The CArdiovascular Risk Evaluation in Men With Prostate Cancer Study (CARE-PC): Initial Pilot Feasibility Study to Assess Patient Awareness and Risk Mitigation
Brief Title: The CArdiovascular Risk Evaluation in Men With Prostate Cancer Study (CARE-PC) Pilot Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Narayan (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor-Investigator, Vivek Narayan, Principal Investigator, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 07823; 853844 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men With Prostate Cancer Planned for Receiving ADT (Other): Men with prostate cancer > 18 years of age who are currently receiving or will be receiving treatment with ≥ 6 months of systemic androgen deprivation therapy (ADT).
  Interventions: Behavioral: CARE-PC Web-Based Application

INTERVENTIONS:
Behavioral: CARE-PC Web-Based Application — The CARE-PC app is a pragmatic, patient-oriented, web-based application that enables the education of patients regarding cardiovascular (CV) risks and collects CV and prostate cancer-related risk variables and CV care access data from prostate cancer patients receiving ADT.

SUMMARY:
The overarching goal of this trial is to develop mechanisms to improve cardiovascular care among such prostate cancer patients receiving ADT by increasing patient awareness of individualized cardiovascular risk estimates and mitigation opportunities. Patients will be given access to a web-based quality improvement tool to educate patients of cardiovascular risks in prostate cancer and to inform them of their individualized, estimated cardiovascular risk and guideline-based risk mitigation recommendations.

The study will assess the feasibility of this web-based application as a cardiovascular education tool for patients with prostate cancer.

The study will also evaluate if completion of the web-based tool improves cardiovascular care access and risk mitigation for patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men with prostate cancer > 18 years of age who are currently receiving or will be receiving treatment with ≥ 6 months of ADT
* Patients must be able to read and understand English.

Exclusion Criteria: n/a

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
CARE-PC Web-Based Application Completion Rate | 18 months
  Completion rate measured as the proportion of participants successfully completing the web-based application out of the total number of subjects approached.

SECONDARY OUTCOMES:
Patient acceptance and perception of the web-based application | 18 months
  Acceptance/perception measured by brief embedded survey following participation in the web-based application
Percent accuracy of patient-derived CV- and prostate cancer-related data elements | 18 months
  Accuracy assessed through parallel medical chart review by cardiology and oncology clinicians
Prevalence of CV risk factors/disease at the time of CARE-PC web-based application participation | 18 months
  Prevalence assessed through parallel medical chart review by cardiology and oncology clinicians
Proportion of participants with current cardiologist involvement in CV care at the time of web-based application participation | 18 months
  Patient reported cardiologist involvement via CARE-PC application at time of application survey completion
Proportion of participants engaging in CV care within 6 months of CARE-PC web application participation | 18 months
  CV care engagement assessed through medical chart review by investigators within 6 months post-application survey completion
Proportion of participants having changes in CV risk-reducing medications within 6 months of CARE-PC application participation. | 18 months
  Proportion of participants having changes in CV risk-reducing medications assessed through parallel medical chart review by cardiology and oncology clinicians within 6 months post-application survey completion

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Narayan, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT06064149/Prot_SAP_000.pdf